CLINICAL TRIAL: NCT05764330
Title: Weight Loss Interventions to Reduce Cancer Progression in Prostate Cancer Patients Under Active Surveillance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I-2980822; NCI-2023-01092 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-2980822 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2023-02-21; First posted 2023-03-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Diet Therapy; Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (CER) (Active Comparator): Patients undergo CER intervention consisting of remote lesson containing information and behavioral strategies about weight loss, session with study interventionist to review lessons, and self-monitoring of body weight. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Dietary Intervention
- Arm II (IF) (Experimental): Patients undergo IF intervention consisting of remote lesson containing information and behavioral strategies about fasting, session with study interventionist to review lessons, and self-monitoring of body weight. Patients also undergo fasting 2 days per week and eat according to the NCI guidelines the remaining 5 days. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Dietary Intervention; Behavioral: Fasting

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Dietary Intervention — Undergo CER intervention
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm I (CER)
Other: Dietary Intervention — Undergo IF intervention
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm II (IF)
Behavioral: Fasting — Undergo fasting
  Other Names: Fast
  Arms: Arm II (IF)

SUMMARY:
This clinical trial examines weight loss interventions in reducing cancer progression in prostate cancer patients under active surveillance. Intensive lifestyle interventions that recommend modest reductions in daily caloric intake (i.e. continuous calorie energy reduction [CER]) are the gold-standard for weight loss, and have been tested in cancer survivors, including prostate cancer patients. However, few interventions have been developed for low-risk prostate cancer patients on active surveillance. Intermittent fasting (IF) may be superior to CER in the context of prostate cancer progression given its dual role in weight loss and metabolic switching from the use of glucose as a fuel source to the use of fatty acids and ketone bodies. This study may help researchers determine which weight loss strategies can reduce their risk of prostate cancer recurrence, and other negative health effects of being overweight or obese.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop two evidence-based behavioral weight loss intervention programs (IF and CER) with a goal to cause weight loss in prostate cancer (PCa) patients on active surveillance (AS).

II. Determine the initial comparative effectiveness of two intervention programs (IF and CER) on weight loss and PCa progression outcomes.

SECONDARY OBJECTIVE:

I. Compare the effects of the interventions on biomarkers underlying obesity and PCa to provide mechanistic insights and potential surrogate biomarkers for PCa prognosis.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo the CER intervention consisting of remote lessons containing information and behavioral strategies about weight loss, session with study interventionist to review lessons, and self-monitoring of body weight, physical activity and dietary intake. Patients also undergo collection of blood samples throughout the trial.

ARM II: Patients undergo IF intervention consisting of remote lesson containing information and behavioral strategies about fasting, session with study interventionist to review lessons, and self-monitoring of fasting. Patients will undergo fasting 2 days per week and eat according to the National Cancer Institute (NCI) guidelines the remaining 5 days. Patients also undergo collection of blood samples throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older (no upper limit)
* Body mass index (BMI) >= 25 kg/m^2
* English speaking
* Not currently on weight loss medications
* Prostate cancer patients who are under active surveillance (including observation) and actively followed at Roswell Park
* Not under active treatment for other cancer diagnosis
* Free of medical problems that might contraindicate participation in a behavioral weight reduction program containing an exercise component
* Has not lost at least 10% of their body weight in the last 6 months
* Has not had bariatric surgery in the last 10 years
* Able to walk unassisted and continuously for 10 minutes
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Unable to consent
* Unwilling or unable to follow protocol requirements
* Unable to complete study measures in English
* Adults who have had a myocardial infarction (heart attack) or stroke without medical clearance from their primary care physician to participate in the study
* Adults who currently have type 1 or type 2 diabetes without medical clearance from their primary care physician to participate in the study
* History of partial or radical prostatectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Body weight | Up to 6 months
  Weight will be measured using a body composition monitor.
Changes in prostate cancer (PCa) progression | Up to 6 months
  Will assess changes in PCa progression indicated by serum prostate specific antigen (PSA) doubling time, and biopsy tumor upgrading and/or upstaging if required clinically, between the timepoints prior and post to the intervention. The timing of the intervention and data collection visits will be scheduled to correspond with the PCa patient's regular management check-up with their physician to allow their scheduled PSA test fall within at least a 6-month time window. For patients if prostate biopsy per clinical guidance is scheduled within 6 months after the intervention, the results from the biopsy post to the intervention as well as the nearest biopsy prior to the intervention will be requested. PSA test results (level and doubling time) and pathology reports on biopsies tissues (stage and grade) will be requested from the Biomedical Research Informatics Shared Resource for both baseline and follow-up visits and defined based on clinical criteria.

SECONDARY OUTCOMES:
Dietary intake | Up to 6 months
  Will confirm the extent changes in body weight are due to changes in caloric intake. Dietary intake will be assessed by the interview administered Nutrition Data System for Research.
Physical activity | Up to 6 months
  Will be assessed using the Paffenbarger Physical Activity Questionnaire (PAQ). The PAQ provides an estimate of calories expended per week in overall leisure time activity and in activities of light (5 kcal/min), medium (7.5 kcal/min) and high (19 kcal/min) intensity.
Change from baseline in Prostate Cancer related biomarkers | Up to 6 months
  Correlation of weight loss and PCa biomarkers.
Change in Urinary functions | Up to 6 months
  urinary function changes will be tracked using a validated questionnaire, the International Prostate Symptom Score
Improvement of Quality of life | Up to 6 months
  Self-reported outcomes routinely collected at each follow up clinic visit using validated questionnaire - UCLA PCI for quality of life.The UCLA PCI domain is scored on a scale of 0-100 points with higher values representing better outcomes.
Change in Sexual functions | Up to 6 months
  Sexual health inventory for men (SHIM). The total score is obtained by adding all five item scores, and can range from 5 to 25. Higher scores indicate higher level of sexual function and less erectile dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeary, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States